CLINICAL TRIAL: NCT02223455
Title: Building an Optimal Hand Hygiene Bundle: A Mixed Methods Approach
Brief Title: Building an Optimal Hand Hygiene Bundle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: CRE 12-289
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Hand Hygiene; Health Care Associated Infection; Compliance
Keywords: Methicillin-resistant Staphylococcus aureus (MRSA); Infection Control (IC); Hospital-associated infections (HAI); Hand Hygiene (HH); Compliance; Health Care Workers (HCWs)
MeSH Terms: conditions — Cross Infection; Patient Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single Hand Hygiene Sign (Placebo Comparator): Wards/units in this arm of the study will have the same hand hygiene sign posted by the hand sanitizer dispensers outside each patient room. The sign will not change.
  Interventions: Other: Hand Hygiene Signs
- Hand Hygiene Signs Changed Monthly (Active Comparator): Intervention: Hand Hygiene Signs Changed Monthly Hand hygiene signs will be changed monthly on wards/units randomized to this arm of the study. Signs will be posted by the hand hygiene sanitizer outside each patient room.
  Interventions: Other: Hand Hygiene Signs
- Hand Hygiene Signs Changed Weekly (Active Comparator): Intervention: Hand Hygiene Signs Changed Weekly Hand hygiene signs will be changed weekly on wards/units randomized to this arm of the study. Signs will be posted by the hand hygiene sanitizer outside each patient room.
  Interventions: Other: Hand Hygiene Signs

INTERVENTIONS:
Other: Hand Hygiene Signs — Hand hygiene signs will not be changed (control) or change weekly/monthly on wards/units randomized to each of these study arms. Signs will be posted by the hand hygiene sanitizer outside each patient room.

SUMMARY:
Hand hygiene is the single most effective practice in preventing the spread of hospital-acquired infections. Despite the strength of the evidence, hospital staff continue to sanitize their hands less than half of the time required by guidelines. Effective interventions are needed to improve hand hygiene compliance rates among hospital staff, but most are of poor quality and do not examine the specific effects of individual interventions. This study will build a "bundle" of three hand hygiene interventions using a research design that allows for the effectiveness of each intervention to be measured individually and combined.

DETAILED DESCRIPTION:
The two specific aims and associated hypotheses of CREATE Project 2 include:

1. Identify combinations of hand-hygiene intervention strategies that optimize hand-hygiene compliance and that could form an evidence-based hand-hygiene bundle for Veterans Health Administration (VHA) implementation.

   Hypothesis 1: Combinations of interventions will increase compliance rates more than single interventions.

   Aim 1 will entail a 30-month cluster-randomized controlled trial that will sequentially test three individual hand-hygiene interventions - hand-hygiene point-of-use reminder signs to serve as an environmental cue to action, individual hand sanitizers, and health care worker hand cultures - to identify an optimal combination of interventions to increase hand-hygiene compliance. The trial will be conducted in 59 hospital units in 10 VA hospitals in order to test the efficacy of individual and then sequentially added interventions to determine their incremental impact on hand-hygiene compliance.

   The focus for this clinical trial will be on Aim 1--Single Hand Hygiene Sign changes.
2. Identify institutional, organizational, ward/ICU, and individual level facilitators and barriers to implementing hand-hygiene interventions.

Hypothesis 2: Facilitators and barriers will pattern around contextual factors such as level of leadership support and organization of infection control programs.

Aim 2 will entail a qualitative process evaluation that includes site visits to purposefully selected sites, semi-structured interviews, and observations to examine barriers and facilitators to the interventions and develop contextual insight for implementing and scaling-up the intervention at additional sites as a national initiative.

ELIGIBILITY:
Inclusion Criteria:

* Wards/units at 10 VA medical centers: hand hygiene observations of healthcare works on these wards/units

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather S Reisinger, PhD, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (10):
- United States (10):
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
As requested
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: August 2020 for 7 years
Access Criteria: IRB and VA Research and Development approval of protocol for sharing

REFERENCES:
- [Derived] Vander Weg MW, Perencevich EN, O'Shea AMJ, Jones MP, Vaughan Sarrazin MS, Franciscus CL, Goedken CC, Baracco GJ, Bradley SF, Cadena J, Forrest GN, Gupta K, Morgan DJ, Rubin MA, Thurn J, Bittner MJ, Reisinger HS. Effect of Frequency of Changing Point-of-Use Reminder Signs on Health Care Worker Hand Hygiene Adherence: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2019 Oct 2;2(10):e1913823. doi: 10.1001/jamanetworkopen.2019.13823. PMID 31642930

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: inpatient wards/units
Period: Overall Study
Arm/Group | Single Hand Hygiene Sign | Hand Hygiene Signs Changed Monthly | Hand Hygiene Signs Changed Weekly
Started | NA; 19 inpatient wards/units (Participant level data not collected.) | NA; 19 inpatient wards/units (Participant level data not collected.) | NA; 20 inpatient wards/units (Participant level data not collected.)
Completed | NA; 19 inpatient wards/units (Participant level data not collected.) | NA; 19 inpatient wards/units (Participant level data not collected.) | NA; 20 inpatient wards/units (Participant level data not collected.)
Not Completed | NA; 0 inpatient wards/units | NA; 0 inpatient wards/units | NA; 0 inpatient wards/units

BASELINE CHARACTERISTICS:
Population: This study is a cluster randomized control trial. Outcomes are measured by unit/ward not individual participant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Hand Hygiene Sign | Hand Hygiene Signs Changed Monthly | Hand Hygiene Signs Changed Weekly | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Continuous — We did not collect age at a participant level. Data are aggregated at the unit level.
Sex: Female, Male — We did not collect sex at a participant level. Data are aggregated at the unit level
Region of Enrollment [unit: ward/unit]

OUTCOME MEASURES:

1. Primary Outcome: Hand Hygiene Compliance
Description: Hand hygiene compliance is the primary outcome measure. Compliance rates will be determined using the same methods of direct observation of HCWs developed by Dr. Perencevich for his VA Health Services Research & Development (HSR&D) funded study (IIR 09-099). Compliance will be collected monthly throughout the project for each of the 59 units.
Time Frame: phase 1 (7-12 months) thru phase 3 (19-21 months)
Population: Entry and exit HH compliance were calculated for units in each treatment group. Crude (unadjusted) change in HH compliance from baseline to follow-up was assessed for each intervention group using Fisher's exact test.
Measure: Mean (95% Confidence Interval); unit: percentage of change in HH compliance
Units Other Than Participants: inpatient wards/units
Groups:
- Single Hand Hygiene Sign: Wards/units in this arm of the study will have the same hand hygiene sign posted by the hand sanitizer dispensers outside each patient room. The sign will not change.
  Hand Hygiene Compliance Signs: Hand hygiene signs will not be changed (control) or change weekly/monthly on wards/units randomized to each of these study arms. Signs will be posted by the hand hygiene sanitizer outside each patient room.
- Hand Hygiene Signs Changed Monthly: Hand hygiene signs will be changed monthly on wards/units randomized to this arm of the study. Signs will be posted by the hand hygiene sanitizer outside each patient room.
  Hand Hygiene Compliance Signs: Hand hygiene signs will not be changed (control) or change weekly/monthly on wards/units randomized to each of these study arms. Signs will be posted by the hand hygiene sanitizer outside each patient room.
- Hand Hygiene Signs Changed Weekly: Hand hygiene signs will be changed weekly on wards/units randomized to this arm of the study. Signs will be posted by the hand hygiene sanitizer outside each patient room.
  Hand Hygiene Compliance Signs: Hand hygiene signs will not be changed (control) or change weekly/monthly on wards/units randomized to each of these study arms. Signs will be posted by the hand hygiene sanitizer outside each patient room.
Arm/Group | Single Hand Hygiene Sign | Hand Hygiene Signs Changed Monthly | Hand Hygiene Signs Changed Weekly
Number analyzed (Participants) | NA | NA | NA
Number analyzed (inpatient wards/units) | 19 | 19 | 20
percentage of change in HH compliance
  Room Entry | -0.4 [-20.5 to 23.0] | 1.8 [-21.5 to 29.7] | -1.3 [-17.9 to 17.4]
  Room Exit | -3.7 [-16.4 to 10.2] | -5.2 [-16.2 to 6.7] | 1.8 [-11.1 to 16.1]

ADVERSE EVENTS:
Description: Adverse Events were not collected because of the nature of the trial - no individual level data collected.
Arm/Group | Single Hand Hygiene Sign | Hand Hygiene Signs Changed Monthly | Hand Hygiene Signs Changed Weekly
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No